CLINICAL TRIAL: NCT03184558
Title: A Phase II, Multi Centre Study of BGB324 in Combination With Pembrolizumab in Patients With Previously Treated, Locally Advanced and Unresectable or Metastatic Triple Negative Breast Cancer (TNBC) or Triple Negative Inflammatory Breast Cancer (TN-IBC)
Brief Title: Bemcentinib (BGB324) in Combination With Pembrolizumab in Patients With TNBC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on planned futility assessment
Sponsor: BerGenBio ASA (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGBC007; MK-3475 PN530 (Other: MSD); 2016-003608-30 (EudraCT Number)
Record Dates: First submitted 2017-05-30; First posted 2017-06-12 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Triple Negative Breast Cancer; Inflammatory Breast Cancer Stage IV
Keywords: bemcentinib; TNBC; pembrolizumab; Keytruda; BGB324
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — bemcentinib; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Extension to Simon's 2-stage design allowing termination at the end of Stage 1 for either futility or efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bemcentinib (BGB324) + pembrolizumab (Experimental): Participants received Bemcentinib (BGB324) capsules orally once daily as a loading dose of 400 milligram (mg) on Days 1, 2, and 3. A dose of 200 mg pembrolizumab was given by intravenous infusion over 30 minutes every 3 weeks in all participants. Dosing of both drugs commenced on Day 1. On days when both BGB324 and pembrolizumab were given, pembrolizumab was given first and participants were observed for 1 hour after the end of infusion before BGB324 was administered. From Day 4 onward, participants received a daily maintenance dose of 200 mg along with Pembrolizumab 200 mg intravenous (IV) infusion over 30 minutes every 3 weeks until disease progression, until an unacceptable toxicity occurred that required treatment withdrawal or withdrawal of consent or until 106 weeks had passed.
  Interventions: Drug: Bemcentinib; pembrolizumab

INTERVENTIONS:
Drug: Bemcentinib; pembrolizumab — Bemcentinib is a selective Axl kinase inhibitor; pembrolizumab is a programmed death receptor-1 (PD-1) inhibitor.
  Other Names: BGB324; Keytruda

SUMMARY:
This is an open label, single arm, multi-centre phase II study to assess the anti-tumour activity and safety of bemcentinib (BGB324) in combination with pembrolizumab in participants with previously treated, locally advanced and unresectable, or metastatic TNBC or TN-IBC. The primary objective is objective response rate.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed informed consent.
2. Male and non-pregnant females who are aged 18 years or older at the time of provision of informed consent.
3. Histopathologically or cytologically documented TNBC or TN-IBC. Tumors must have been confirmed negative for ER and partial response (PR) by immunohistochemistry (IHC) (<1% positive tumor nuclei, as per ASCO-CAP guideline recommendations) and negative for human epidermal growth factor receptor 2 (HER2) by IHC or fluorescent or chromogenic in situ hybridization (FISH or CISH). Patients with equivocal HER2 results by IHC should have their negativity status confirmed by FISH.
4. Locally advanced and unresectable or metastatic TNBC or triple negative inflammatory breast cancer.
5. Received one or more prior therapies for TNBC or inflammatory breast cancer in the metastatic setting, and prior treatment (metastatic or (neo) adjuvant) must have included a prior taxane and/or anthracycline-based therapy.
6. Has measurable disease as defined by RECIST 1.1 on computed tomography (CT) or magnetic resonance imaging (MRI) and as determined by the site study team. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. Provision of suitable tumor tissue for the analysis of Axl kinase expression and PD-L1 expression.
8. Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
9. Life expectancy of at least 3 months.
10. Adequate organ function confirmed at Screening and within 10 days of initiating treatment, as evidenced by:

    * Platelet count ≥100,000 /mm3;
    * Hemoglobin ≥9.0 g/dL (≥5.6 mmol/L);.
    * Absolute neutrophil count (ANC) >1,500 /mm^3;
    * Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤2.5 times the upper limit of normal (ULN), or ≤5 times the ULN for patients with liver metastases;
    * Total bilirubin ≤1.5 times the ULN, or direct bilirubin <ULN for patients with total bilirubin levels >1.5xULN;
    * Creatinine ≤1.5 times the ULN and calculated creatinine clearance >60 mL/min (by Cockcroft Gault formula);
    * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 times the ULN and Activated Partial Thromboplastin Time (aPTT) ≤1.5 times the ULN. Note: If patient is receiving anticoagulant therapy, then PT or PTT must be within therapeutic range of intended use of anticoagulants;
    * Lactate dehydrogenase (LDH) ≤2.5 times the ULN.
11. Female patients of childbearing potential must have a negative pregnancy test (either urine or serum pregnancy test) within 72 hours prior to the first dose of study treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Have resolution of toxic effect(s) of the most recent prior chemotherapy to Grade 1 or less (except alopecia). If the patient received major surgery or radiation therapy of >30 Gy, they must have recovered from the toxicity and/or complications from the intervention.
13. Patients of reproductive potential must be willing to practice highly effective methods of contraception throughout the study and for 120 days after the last dose of study medication. Abstinence is acceptable if this is the usual lifestyle of the patient.

Exclusion Criteria:

1. Has disease that is suitable for local therapy administered with curative intent.
2. More than 3 previous lines of therapy in the metastatic setting.
3. Has received prior therapy with an immunomodulatory agent.
4. Has a known additional malignancy that is progressing or requires active treatment. Note: Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
5. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
6. History of the following cardiac conditions:

   * Congestive cardiac failure of >Grade II severity according to the New York Heart Association (NYHA);
   * Ischemic cardiac event including myocardial infarction within 3 months prior to first dose;
   * Uncontrolled cardiac disease, including unstable angina, uncontrolled hypertension (i.e. sustained systolic BP >160 mmHg or diastolic BP >90 mmHg), or need to change medication due to lack of disease control within 6 weeks prior to the provision of consent;
   * History or presence of sustained bradycardia (≤55 BPM), left bundle branch block, cardiac pacemaker or ventricular arrhythmia. Note: Patients with a supraventricular arrhythmia requiring medical treatment, but with a normal ventricular rate are eligible;
   * Family history of long QTc syndrome; personal history of long QTc syndrome or previous drug-induced QTc prolongation of at least Grade 3 (QTc >500 ms).
7. Abnormal left ventricular ejection fraction on echocardiography or Multi Gated Acquisition Scan (MUGA) (less than the lower limit of normal for a patient of that age at the treating institution or <45%, whichever is lower).
8. Current treatment with any agent known to cause Torsades de Pointes which cannot be discontinued at least five half-lives or two weeks prior to the first dose of study treatment.
9. Screening 12-lead ECG with a measurable QTc interval according to Fridericia's correction >450 ms.
10. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study treatment.
11. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤Grade 1 or at baseline) from AEs due to a previously administered agent.
12. Received an anti-cancer monoclonal antibody (mAb) within 4 weeks prior to the first dose of study treatment or who has not recovered (i.e. ≤Grade 1 or baseline) from AEs due to agents administered more than 4 weeks earlier.
13. Major surgery within 28 days prior to start of study treatment and failure to have recovered adequately from the toxicity and/or complications from the intervention prior to the first dose of study treatment.
14. Received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte-colony stimulating factor [G-CSF], Granulocyte-macrophage colony-stimulating factor [GM-CSF] or recombinant erythropoetin) within 4 weeks prior to the first dose of study treatment.
15. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
16. Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
17. Known history of human immunodeficiency virus (HIV 1/2 antibodies)
18. Has known active infection with Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., Hepatitis C virus (HCV) RNA (qualitative) is detected).
19. Has received a live-virus vaccination within 30 days of planned treatment start. Note: Seasonal flu vaccines that do not contain live virus are permitted.
20. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
21. Has a history of interstitial lung disease.
22. Inability to swallow or tolerate oral medication.
23. Existing gastrointestinal disease affecting drug absorption such as celiac disease or Crohn's disease, or previous bowel resection which is considered to be clinically significant or could interfere with absorption.
24. Known lactose intolerance.
25. Requires vitamin K antagonists. Note: Patients receiving low doses prescribed to maintain the patency of venous access devices may be included. Factor Xa antagonists are permitted.
26. Treatment with any of the following: histamine receptor 2 inhibitors, proton pump inhibitors or antacids within 7 days of start of study treatment.
27. Treatment with any medication which is predominantly metabolized by CYP3A4 and has a narrow therapeutic index.
28. Known severe hypersensitivity (≥Grade 3) to bemcentinib, pembrolizumab, and/or any of their excipients.
29. Has an active infection requiring systemic therapy (apart from cutaneous infections).
30. Has a history or current evidence of any condition, therapy, or laboratory abnormality that, in the opinion of the Investigator, might confound the results of the trial, interfere with the patient's participation and compliance in the trial, or means it is not in the best interests of the patient to participate.
31. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting from Screening through to 120 days after the last dose of study treatment.
32. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (5):
  - City of Hope Cancer Center, Duarte, California
  - Sharp memorial Hospital, 7901 Frost Street,, San Diego, California
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Magee-Womens Hospital, UPMC Cancer Pavilion, Pittsburgh, Pennsylvania
- Haukeland University Hospital, Bergen, Norway
- Spain (7):
  - University General Hospital of Alicante, Alicante
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Germans Trias i Pujol - Institut Catala d'Oncologia, Barcelona
  - Hospital Universitario Amau de Vilanova de Lieda, Servicio de Oncologia, Lleida
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Imperial College Healthcare NHS Trust, Charing Cross Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals, City Campus, Hucknall Road, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification [text, tables, figures and appendices].
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Proposal should be directed to HYPERLINK "mailto:clinical@bergenbio.com" clinical@bergenbio.com. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 29 participants were enrolled and received study medication in this study.
Groups:
- Bemcentinib + Pembrolizumab: Participants received Bemcentinib (BGB324) capsules orally once daily as a loading dose of 400 milligram (mg) on Days 1, 2, and 3. A dose of 200 mg pembrolizumab was given by intravenous infusion over 30 minutes every 3 weeks in all participants. Dosing of both drugs commenced on Day 1. On days when both BGB324 and pembrolizumab were given, pembrolizumab was given first and participants were observed for 1 hour after the end of infusion before BGB324 was administered. From Day 4 onward, participants received a daily maintenance dose of 200 mg along with Pembrolizumab 200 mg intravenous (IV) infusion over 30 minutes every 3 weeks until disease progression, until an unacceptable toxicity occurred that required treatment withdrawal or withdrawal of consent or until 106 weeks had passed.
Period: Overall Study
Arm/Group | Bemcentinib + Pembrolizumab
Started | 29
Completed | 0
Not Completed | 29
Not completed — Withdrawal by Subject | 2
Not completed — Death | 16
Not completed — Lost to Follow-up | 2
Not completed — Other | 9

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who were enrolled in the study and who received at least 1 dose of study product (BGB324 and/or pembrolizumab).
Arm/Group | Bemcentinib + Pembrolizumab
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of evaluable participants who had at least one confirmed overall response of complete response (CR) or partial response (PR) according to the modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. CR: Disappearance of all target lesions (TLs) since baseline, any pathological lymph nodes selected as TLs must have a reduction in short axis to less than (<) 10 millimeter (mm). PR: At least a 30 percent decrease in the sum of the diameters of TLs, taking as reference the baseline sum of diameters.
Time Frame: Until disease progression or death or withdrawal of consent whichever comes first, up to end of study (Up to 1 year)
Population: The Evaluable analysis set (EAS) included all evaluable participants who had received at least 1 combination dose of pembrolizumab and bemcentinib and who had measurable disease at entry, as determined by the investigator site assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Bemcentinib + Pembrolizumab
Number analyzed (Participants) | 29
percentage of participants | 0

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the date of first documented response until date of documented progression or death in the absence of disease progression (PD); the end of response should coincide with the date of progression or death from any cause. PD per modified RECIST 1.1 defined as: at least a 20 percent increase in the sum of diameters of TLs and an absolute increase of at least 5 mm, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Until disease progression or death or withdrawal of consent whichever comes first, up to end of study (Up to 1 year)
Population: Analysis performed on participants in EAS who had an objective response. DOR could not be calculated as none of the participants had an objective response.
Arm/Group | Bemcentinib + Pembrolizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with a confirmed CR, PR, or stable disease (SD). CR: Disappearance of all target lesions (TLs) since baseline, any pathological lymph nodes selected as TLs must have a reduction in short axis to < 10 mm. PR: At least a 30 percent decrease in the sum of the diameters of TLs, taking as reference the baseline sum of diameters. SD per modified RECIST 1.1 defined as: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Until disease progression or death or withdrawal of consent whichever comes first, up to end of study (Up to 1 year)
Population: The evaluable analysis set included all evaluable participants who had received at least 1 combination dose of pembrolizumab and bemcentinib and who had measurable disease at entry, as determined by the investigator site assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Bemcentinib + Pembrolizumab
Number analyzed (Participants) | 29
percentage of participants | 3.4

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the duration from start of treatment until the date of radiological disease progression (the date on which the confirmed progression was initially observed) or the date of death (regardless of cause of death), whichever was earlier.
Time Frame: Until disease progression or death or withdrawal of consent whichever comes first, up to end of study (Up to 1 year)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Bemcentinib + Pembrolizumab
Number analyzed (Participants) | 29
Weeks | 13.1 [12.4 to 18.3]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first dose of study treatment until the date of death (from any cause and irrespective of any subsequent anti-cancer treatment given).
Time Frame: Until disease progression or death or withdrawal of consent whichever comes first, up to end of study (Up to 1 year)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Bemcentinib + Pembrolizumab
Number analyzed (Participants) | 29
Weeks | 32.0 [13.6 to 37.1]

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: The safety set included all participants who were enrolled in the study and who received at least 1 dose of study product (bemcentinib and/or pembrolizumab).
Arm/Group | Bemcentinib + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 16/29
Serious Adverse Events (participants affected / at risk) | 22/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bemcentinib + Pembrolizumab (N=29)
Pyrexia (General disorders) | 5
Adverse drug reaction (General disorders) | 1
Face oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 4
Transaminases increased (Investigations) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bemcentinib + Pembrolizumab (N=29)
Fatigue (General disorders) | 12
Pyrexia (General disorders) | 6
Pain (General disorders) | 3
Oedema peripheral (General disorders) | 2
Influenza like illness (General disorders) | 3
Axillary pain (General disorders) | 2
Chills (General disorders) | 2
Face oedema (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 6
Abdominal distension (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 3
Aspartate aminotransferase increased (Investigations) | 9
Alanine aminotransferase increased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 5
Electrocardiogram QT prolonged (Investigations) | 4
White blood cell count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Tremor (Nervous system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Oral candidiasis (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hot flush (Vascular disorders) | 3
Hypotension (Vascular disorders) | 2
Insomnia (Psychiatric disorders) | 2
Asthenia (General disorders) | 1
Suprapubic pain (General disorders) | 1
Chest pain (General disorders) | 1
Facial pain (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Paraesthesia oral (Gastrointestinal disorders) | 1
Blood magnesium decreased (Investigations) | 1
Blood thyroid stimulating hormone decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Tri-iodothyronine free decreased (Investigations) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Aphasia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hemiparaesthesia (Nervous system disorders) | 1
Movement disorder (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Conjunctivitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Affect lability (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

LIMITATIONS AND CAVEATS:
None of the participants achieved CR or PR. As there were no responses, the study was terminated. It was planned to terminate the trial in favor of the null hypothesis of futility when 5 or fewer responses were observed in 28 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT03184558/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT03184558/SAP_001.pdf